CLINICAL TRIAL: NCT07048184
Title: Sarcoma Surgery Wound Complications Comparing Usual Versus Negative Pressure Dressing: a Randomised Phase II Trial
Brief Title: Sarcoma Surgery Wound Complications Comparing Usual Versus Negative Pressure Dressing
Acronym: SUNDIAL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Solventum (Industry); Sarcoma UK (Unknown); CRUK Trials unit Glasgow (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN23ON401
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Sarcoma; Negative Pressure Therapy; Wound Complication
Keywords: Sarcoma; Surgery; Wound Complication; Negative Pressure Wound Therapy; NPWT; Dressing; Tumour Resection
MeSH Terms: conditions — Sarcoma | interventions — Negative-Pressure Wound Therapy; Bandages

STUDY DESIGN:
Masking Description: This study will be fully unblinded due to the nature of the wound dressings used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Absorbent Dressing (Active Comparator): Standard Absorbent Dressings for wound closure
  Interventions: Device: Standard Absorbent Dressings
- Negative Pressure Wound Therapy Dressing (Experimental): NPWT Dressings will be used for wound closure
  Interventions: Device: Negative Pressure Wound Therapy (NPWT) Dressings

INTERVENTIONS:
Device: Negative Pressure Wound Therapy (NPWT) Dressings — During wound closure, skin glue is not permitted as this interferes with the NPWT suction mechanism. The NPWT is a mesh-based dressing that will be applied following the transparent occlusive dressing as per the manufacturer's instructions. Patients assigned to NPWT will have their dressing connected to a suction device (ActiV.A.C.®, KCI) providing a constant negative pressure of 125mmHg and left in situ for between 5 and 7 days. The dressings and suction device are all CE-marked medical devices that are being used within their intended usage.
  Arms: Negative Pressure Wound Therapy Dressing
Device: Standard Absorbent Dressings — The wound will be closed as per the standard surgical technique and the operating surgeon's preference. Following wound closure of sarcoma tumour resection, standard absorbent dressing will be applied as per local protocols and the pre-op plan
  Arms: Standard Absorbent Dressing

SUMMARY:
To compare the differences in clinical outcomes and health economics between standard absorbent dressings versus Negative Pressure Wound Therapy dressings following the surgical resection of sarcoma tumours.

DETAILED DESCRIPTION:
The investigators propose to undertake a randomised controlled trial comparing standard absorbent dressings with Negative Pressure Wound Therapy (NPWT) dressings in the wound management following resection of sarcoma tumours. By using, NPWT in sarcoma patients the investigators aim to reduce the number of patients experiencing wound complications compared to those who receive standard absorbent dressings. 94 participants will be recruited over 12 months and randomised in a 1:1 ratio to receive either the standard or NPWT dressings. The primary aim will be to determine whether there is a clinically significant difference in wound complications between standard dressings and NPWT dressings over a four-month post-op period. The investigators will assess the patient's wound for signs of infection, dehiscence and other potential complications, and document the incidence and severity of complications. Researchers will also collect the Musculoskeletal Tumour Society Score (MSTS) and Toronto Extremity Salvage Score (TESS) at pre-op and 4 months post-op to understand how the dressings may have impacted function following recovery. In addition, health economic data will also be captured in the form for ED-5D-5L and questionnaires that will focus on the economic impact of surgery and potential wound complications on a patient return to work.

Wound complications following sarcoma tumour surgery can be traumatic for patients during their recovery and postpone subsequent chemotherapy treatments, as well as being an expensive burden to the NHS. NPWT dressings may potentially offer benefits to both patients and the NHS yet there is insufficient data available to support widespread use of this product in sarcoma patients. It is the investigators belief that NPWT is used because anecdotally it is believed to be better than standard absorbent dressings. However, there is a clear lack of robust evidence to support this idea, and the investigator aim to address this by undertaking this study..

ELIGIBILITY:
Inclusion Criteria:

* Sarcoma of the upper/lower limb or torso requiring wide local excision, planned marginal excision or amputation
* Able to provide informed consent
* Aged 16 years or over
* Able, and willing, to adhere to scheduled trial procedures and visit schedule

Exclusion Criteria:

* Previous surgery to planned surgical field
* Contra-indication to surgical excision of the tumour
* Disseminated malignancy on pre-op radiological imaging
* Post-radiation sarcoma
* Allergy to adhesive dressing
* Subjects who, in the opinion of the PI, will be unable to comply with follow-up

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome: The proportion of patients experiencing wound complications | From surgery to 4 months post-op
  Measured as the proportion of patients with 1 or more wound complications experienced between surgery and the end of post-surgery treatment (4 months after surgery). This will be a binary endpoint for each patient (yes/no).
  Types of wound complication include:
  * Superficial and deep surgical site infections
  * Dehiscence: partial and complete cases
  * Other
Health Economic: The incremental cost per complication avoided | From surgery up to 4 months post-operatively
  Measured using a breadth of health economic data collected during the course of the study to capture the cost of complications, readmissions, EQ5D-5L questionnaire, recovery times and return to work.

SECONDARY OUTCOMES:
Change in EuroQoL-5 Dimensions (EQ-5D-5L) (Patient reported outcome measure of a patients perceptions of their overall health) | Baseline, 28 day post-op and 4 month post-op
  EQ-5D-5L is a validated questionnaire that measures an individual's perception of their overall health. The questionnaire will be completed either face-to-face, via postal questionnaires or via virtual appointments.
  EQ5D-5L has two components, the first is a visual analogue scale where participants rate their overall health one a scale of 0 (worst health state imagined) to 100 (best health state imagined). The second is a descriptive system that assess health across 5 domains (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) each with 5 responses ranging from "no problems" to "extreme problems". These responses provide an individuals health profile that can be converted into a single index score for reporting.
Change in Toronto Extremity Salvage Score (Patient-reported outcome measure of function after limb salvage procedures) | Baseline and 4 months post-operatively
  The Toronto Extremity Salvage Score questionnaire contains 29 items related to various daily tasks and activities. Each item is rated on a 5-point scale, where 1 indicates "impossible to do" and 5 indicates "not at all difficult". The individual item scores are summed, and then the total score is divided by the maximum possible score (based on the number of applicable items) and multiplied by 100 to get a percentage.
Change in Musculoskeletal Tumour Society Score (Clinician-led patient questionnaire used to assess functional outcomes) | Baseline and 4 months pot-operatively
  The Musculoskeletal Tumour Society Score is typically administered by a clinician, who assesses the patient based on the six domains (pain, function, emotional acceptance, support, walking, and gait). Each domain is rated on a scale of 0 to 5, with 0 representing the worst possible outcome and 5 representing the best possible outcome. The individual domain scores are summed to create a total Musculoskeletal Tumour Society Score.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Gupta, MBBS, MRCS, MSc, MPhil, FRCS, Principal Investigator — Department of Trauma and Orthopaedics, Glagow Royal Infirmary, NHS Greater Glasgow and Clyde
Locations (1):
- Glasgow Royal Infirmary, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Semsarzadeh NN, Tadisina KK, Maddox J, Chopra K, Singh DP. Closed Incision Negative-Pressure Therapy Is Associated with Decreased Surgical-Site Infections: A Meta-Analysis. Plast Reconstr Surg. 2015 Sep;136(3):592-602. doi: 10.1097/PRS.0000000000001519. PMID 26313829
- [Background] Bedi M, King DM, DeVries J, Hackbarth DA, Neilson JC. Does Vacuum-assisted Closure Reduce the Risk of Wound Complications in Patients With Lower Extremity Sarcomas Treated With Preoperative Radiation? Clin Orthop Relat Res. 2019 Apr;477(4):768-774. doi: 10.1097/CORR.0000000000000371. PMID 30811365
- [Background] Ouyang Z, Trent S, McCarthy C, Cosker T, Stuart R, Pratap S, Whitwell D, White HB, Tao H, Guo X, Maxime Gibbons CL. The incidence, risk factors and outcomes of wound complications after preoperative radiotherapy and surgery for high grade extremity soft tissue sarcomas: A 14-year retrospective study. Eur J Surg Oncol. 2023 Nov;49(11):107086. doi: 10.1016/j.ejso.2023.107086. Epub 2023 Sep 16. PMID 37741042
- [Background] O'Sullivan B, Davis AM, Turcotte R, Bell R, Catton C, Chabot P, Wunder J, Kandel R, Goddard K, Sadura A, Pater J, Zee B. Preoperative versus postoperative radiotherapy in soft-tissue sarcoma of the limbs: a randomised trial. Lancet. 2002 Jun 29;359(9325):2235-41. doi: 10.1016/S0140-6736(02)09292-9. PMID 12103287
- [Background] Shields DW, Razii N, Doonan J, Mahendra A, Gupta S. Closed incision negative pressure wound therapy versus conventional dressings following soft-tissue sarcoma excision: a prospective, randomized controlled trial. Bone Jt Open. 2021 Dec;2(12):1049-1056. doi: 10.1302/2633-1462.212.BJO-2021-0103.R1. PMID 34905941
- [Background] Nandra R, Hwang N, Matharu GS, Reddy K, Grimer R. One-year mortality in patients with bone and soft tissue sarcomas as an indicator of delay in presentation. Ann R Coll Surg Engl. 2015 Sep;97(6):425-33. doi: 10.1308/003588415X14181254790284. Epub 2015 Aug 14. PMID 26274756
- See also: UK S. Sarcoma Incidence — https://sarcoma.org.uk/about-sarcoma/what-is-sarcoma/sarcoma-incidence/
- See also: EUROQOL. EQ-5D-5L User Guide 2023 — https://euroqol.org/wp-content/uploads/2023/11/EQ-5D-5LUserguide-23-07.pdf.